CLINICAL TRIAL: NCT00168584
Title: Randomised Study of the Impact of Different Doses of Vitamin A on Childhood Morbidity and Mortality
Brief Title: Different Doses of Vitamin A and Childhood Morbidity and Mortality
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91096-2dos02; 91096-02
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-09

CONDITIONS: Mortality; Morbidity
Keywords: Vitamin A; Mortality; Morbidity; Doses; OPV
MeSH Terms: interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
Vitamin A supplementation reduces all-cause mortality. It is therefore given with oral polio vaccine in national campaigns. However, it is not clear which dose is optimal. The two studies that have investigated the impact of different doses of vitamin A have both found that a smaller dose was better than a large dose. We therefore investigated if a smaller dose given with oral polio vaccine gives equal or better effect.

DETAILED DESCRIPTION:
Vitamin A supplementation (VAS) to children above 6 months of age reduces all-cause mortality with 23 %1 to 30 % in low-income countries. WHO recommends VAS at vaccination contacts. The currently recommended doses to be administered every 3-6 months are 100,000 IU for infants between 6 and 11 months of age and 200,000 IU for children 12 months and older. There is no clear evidence that a large dose is better than a small dose, the tendency being the opposite in the two studies of different doses of VAS that have been published so far.

With the global effort to eradicate polio, national immunization days with oral polio vaccine (OPV) offer an additional opportunity to provide vitamin A. In Guinea-Bissau, a combined OPV and VAS campaign took place in November 2002. Given the uncertainty about the best dose of VAS, we aimed to examine whether the dose of vitamin A currently recommended by WHO or half this dose gives a better protection against childhood morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:Between 6 mo and 5 years old and thus eligible for OPV and vitamin A during national immunisation day

-

Exclusion Criteria:Children with overt signs of vitamin A deficiency will not be enrolled in the study, but treated according to the recommendations. -

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5400
Dates: Start 2002-11; Study Completion 2003-08

PRIMARY OUTCOMES:
Mortality
Hospitalisations
Morbidity
Growth

SECONDARY OUTCOMES:
Rotavirus infection

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, DMSc, Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau